CLINICAL TRIAL: NCT02474693
Title: Assessment of the Proportion of Sodium Intake From a Variety of Sources - Salt Sources Study
Brief Title: Salt Sources Study
Status: Completed | Type: Observational
Sponsor: Mary Cogswell (U.S. Federal Agency)
Collaborators: University of Minnesota (Other); University of Birmingham (Other); Stanford University (Other)
Responsible Party: Sponsor-Investigator, Mary Cogswell, Senior Scientist, Centers for Disease Control and Prevention
Organization: Centers for Disease Control and Prevention (U.S. Federal Agency)
Other Study IDs: 0920-0982
Record Dates: First submitted 2015-05-12; First posted 2015-06-18 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Dietary Sources of Sodium Intake

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 24 hour urine samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The Centers for Disease Control and Prevention conducted an observational cross-sectional study to obtain information about the amount of sodium consumed from various sources (including sodium from processed and restaurant foods, sodium inherent in foods, and salt added at the table and during cooking) and to examine variability across population subgroups. Data collection will include an observational component as well as a sub-study designed to refine the accuracy of estimates of total sodium intake and discretionary sodium intake.

Information was collected in three distinct geographic regions: 1) Minneapolis/St. Paul, Minnesota, 2) Birmingham, Alabama, and 3) Palo Alto, California. Over a two-year period, a study center in each location recruited 150 participants (total N=450). Overall, an approximately equal number of adults ages 18-74 years by approximately 10-year age groups in each sex-race group, including whites, blacks, Hispanics, and Asians. A sub-study was conducted among a subgroup of 150 of these participants (50 per site). University of Minnesota serves as a study coordinating center.

DETAILED DESCRIPTION:
The Centers for Disease Control and Prevention conducted an observational cross-sectional study to obtain information about the amount of sodium consumed from various sources (including sodium from processed and restaurant foods, sodium inherent in foods, and salt added at the table and during cooking) and to examine variability across population subgroups. Data collection will include an observational component as well as a sub-study designed to refine the accuracy of estimates of total sodium intake and discretionary sodium intake.

Information was collected in three distinct geographic regions: 1) Minneapolis/St. Paul, Minnesota, 2) Birmingham, Alabama, and 3) Palo Alto, California. Over a two-year period, a study center in each location recruited 150 participants (total N=450). Overall, an approximately equal number of adults ages 18-74 years by approximately 10-year age groups in each sex-race group, including whites, blacks, Hispanics, and Asians. A sub-study was conducted among a subgroup of 150 of these participants (50 per site). University of Minnesota serves as a study coordinating center.

After informed consent and completing a screening process, each participant completed a personal questionnaire, a tap water questionnaire, four 24-hour dietary recalls, and four qualitative food records. In addition, height and weight information on each participant were collected, and each participant collected duplicate portions of their cooking/table salt. A few participants at each site also provided water samples analyzed to produce estimates of the amount of sodium in private sources of tap water.

The Salt Sources Study also included a sub-study to help determine the accuracy of estimates of total sodium intake and discretionary salt intake. About 25 participants at each site used a Study Salt for 11 days instead of their own household salt, provide additional information based on four 24-hour urine collections, four follow-up urine collection questionnaires, and three follow-up questionnaires on Study Salt use. The Study Salt has the same amount of sodium and contains a very small amount of lithium, a metal found in trace amounts in all plants and animals and excreted in urine. Participants are instructed to use the study salt as they would their salt at home and to collect duplicate samples of the amount used at the table and during home cooking. The amount of lithium excreted in the 24-hour urine collection is measured to assess the amount of sodium consumed from discretionary salt use (salt used at the table and during home cooking).

Results from the Salt Sources Study will be used to inform public health strategies to reduce sodium intake, determine if substantial variability in sources of sodium intake exists by social and demographic subgroups, and better inform estimates of salt added at the table used in Healthy People 2020 objectives related to sodium reduction.

ELIGIBILITY:
Inclusion Criteria:

* able to read and speak English, who have a telephone
* live in one of three study sites in the following cities or surrounding geographic areas

  1. Minneapolis, Minnesota
  2. Birmingham, Alabama; Palo Alto, California

Exclusion Criteria:

* pregnant
* breastfeeding
* have diabetes insipidus
* have chronic kidney disease.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A convenience sample of adults aged 18-74 years, able to read and speak English, who have a telephone. Respondents will be excluded if they are pregnant, breastfeeding, have diabetes insipidus, or have chronic kidney disease. Information will be collected from the study participants in three study sites in Minnesota, Alabama, and California.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Sodium intake as assessed through four 24 hour dietary recalls | 11 days
  Four 24-hour dietary recalls and duplicate collection of salt added at the table

SECONDARY OUTCOMES:
Discretionary sodium intake from salt added at the table and during cooking as assessed through duplicate salt collection | 11 days
  Collection of duplicated samples of salt added at the table and during cooking on 24-h diet recall days
Total sodium intake as assessed through laboratory analysis 24-h urine collections | 11 days
  Measured from four 24-hour urine collections in a subset of 150 study participants
Discretionary sodium intake (from salt added at the table or during cooking) assessed from the amount of lithium excreted in 24-hour urine collections. | 11 days
  Measured from 24-hour urine collections in a subset of 150 study participants who used lithium labeled salt at the table and for home cooking in place of their usual salt

CONTACTS AND LOCATIONS:
Overall Officials: Lyn Steffen, PhD, MPH, RD, Principal Investigator — University of Minnesota

IPD SHARING:
Plan to Share IPD: Yes
When data cleaning is completed, data can be obtained through submission of a proposal to the proposal and publication committee through contacting one of the investigators

REFERENCES:
- [Derived] Quader ZS, Zhao L, Harnack LJ, Gardner CD, Shikany JM, Steffen LM, Gillespie C, Moshfegh A, Cogswell ME. Self-Reported Measures of Discretionary Salt Use Accurately Estimated Sodium Intake Overall but not in Certain Subgroups of US Adults from 3 Geographic Regions in the Salt Sources Study. J Nutr. 2019 Sep 1;149(9):1623-1632. doi: 10.1093/jn/nxz110. PMID 31179499
- [Derived] Harnack LJ, Cogswell ME, Shikany JM, Gardner CD, Gillespie C, Loria CM, Zhou X, Yuan K, Steffen LM. Sources of Sodium in US Adults From 3 Geographic Regions. Circulation. 2017 May 9;135(19):1775-1783. doi: 10.1161/CIRCULATIONAHA.116.024446. PMID 28483828
- See also: Study description, data collection forms and questionnaires included on the Office of Management and Budget website — http://www.reginfo.gov/public/do/PRAViewICR?ref_nbr=201306-0920-001